CLINICAL TRIAL: NCT05324410
Title: A Phase I, Randomized, Double-blind, Placebo-controlled Study Evaluating the Safety and Pharmacokinetics of Single and Multiple Ascending Doses of VX-840 in Healthy Subjects
Brief Title: A Phase 1 Dose Escalation Study to Evaluate Safety and Pharmacokinetics (PK) of VX-840 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX21-840-001
Record Dates: First submitted 2022-04-05; First posted 2022-04-12 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: APOL1-mediated Kidney Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: VX-840 (Experimental): Participants will be randomized to receive single dose of one of different dose levels of VX-840.
  Interventions: Drug: VX-840
- Part A: Placebo (Placebo Comparator): Participants will receive placebo matched to VX-840.
  Interventions: Drug: Placebo
- Part B: VX-840 (Experimental): Participants will be randomized to receive multiple doses of one of different dose levels of VX-840. The dose levels will be determined based on the data from Part A.
  Interventions: Drug: VX-840
- Part B: Placebo (Placebo Comparator): Participants will receive placebo matched to VX-840.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VX-840 — Solution for oral administration.
  Arms: Part A: VX-840; Part B: VX-840
Drug: Placebo — Placebo matched to VX-840 for oral administration.
  Arms: Part A: Placebo; Part B: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and PK of single and multiple ascending doses of VX-840 in healthy participants.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Female participants must be of non-childbearing potential
* Body mass index (BMI) of 18.0 to 32.0 kilograms per meter square (kg/m^2)
* A total body weight greater than (>) 50 kg

Key Exclusion Criteria:

* History of febrile illness or other acute illness within 14 days before the first dose of study drug
* Any condition possibly affecting drug absorption

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-11-07 (Actual)

PRIMARY OUTCOMES:
Parts A and B: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to Day 25

SECONDARY OUTCOMES:
Parts A and B: Plasma Concentration of VX-840 Over Time | From Day 1 up to Day 14
Part A: Area Under the Concentration Versus Time Curve From the Time of Dosing Extrapolated to Infinity [AUC(0 - inf)] | From Day 1 up to Day 14
Part B: Area Under the Concentration Versus Time Curve From the Time of Dosing to the Last Measurable Concentration [AUC(0-tlast)] | From Day 1 up to Day 14
Part B: Amount of VX-840 Excreted in the Urine During the Dosing Interval (Ae) | From Day 1 up to Day 14
Part B: Associated Renal Clearance (CLr) of VX-840 | From Day 1 up to Day 14

CONTACTS AND LOCATIONS:
Locations (1):
- ICON Lenexa, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing